CLINICAL TRIAL: NCT02386033
Title: Clinical Efficacy of Subgingivally Delivered Atorvastatin in the Treatment of Mandibular Degree II Furcation Defects: A Randomized Controlled Clinical Trial .
Brief Title: Atorvastatin in the Treatment of Mandibular Degree II Furcation Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and head, department of periodontics, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014AB
Record Dates: First submitted 2014-11-30; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRP plus placebo (Placebo Comparator): SRP was done for all the subjects. Placebo gel was delivered subgingivally into the pocket
  Interventions: Drug: Placebo Gel
- SRP plus Atorvastatin (Active Comparator): SRP was done for all the subjects. Atorvastatin was delivered in the pocket subgingivally
  Interventions: Drug: Atorvastatin (ATV)

INTERVENTIONS:
Drug: Atorvastatin (ATV) — After SRP, ATV gel was delivered subgingivally into the pocket
  Other Names: ATV gel
  Arms: SRP plus Atorvastatin
Drug: Placebo Gel — After SRP, placebo gel was delivered subgingivally into the pocket
  Arms: SRP plus placebo

SUMMARY:
ABSTARCT Background: Atorvastatin is an inhibitor of 3-hydroxy-2-methyl-glutaryl coenzyme A reductase. Lately, it has shown to have anti-inflammatory and bone stimulatory effects. The aim of the current study is to explore the effectiveness of 1.2% atorvastatin (ATV) as an adjunct to scaling and root planning (SRP) in the treatment of mandibular degree II furcation defects.

Method: A total of sixty subjects were randomly assigned to two treatment groups. 1. SRP plus placebo gel 2. SRP plus 1.2% ATV gel. Clinical parameters like probing depth (PD), relative vertical clinical attachment level (RVCAL) , relative horizontal clinical attachment level (RHCAL), modified sulcus bleeding index (mSBI) and site specific plaque index were recorded at baseline and then at 3, 6 and 9 months. The radiological assessment of bone defect fill was done at 6 and 9 months, using a computer-aided software.

DETAILED DESCRIPTION:
Two groups were made. One was delivered with ATV after SRP, the other was delivered with placebo gel after SRP.

ELIGIBILITY:
Inclusion Criteria:

* lower first molars demonstrating a probing pocket depth of 5 mm and horizontal probing depth of 3 mm following phase 1 therapy, with furcation defects (degree II) present bucally in asymptomatic, vital lower first molars, with a furcation radiolucency on a periapical radiograph of the molars.

Exclusion Criteria:

* patients with systemic diseases like cardiovascular disease
* diabetes or HIV infection or on medications like corticosteroids which may impede the healing in periodontal tissues.
* pregnant/lactating females
* tobacco users
* alcoholics
* patients with unsatisfactory oral hygiene (plaque index greater than 1.5)
* teeth having gingival recession, caries involving pulp, intrabony defect present interproximally, grade 2/3 mobility
* Furthermore, patients allergic to ATV or other statins or those taking ATV/other statins systemically were excluded.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
amount of bone fill | baseline to 9 months

SECONDARY OUTCOMES:
change in Relative vertical clinical attachment level | baseline to 9 months
change in RHCAL (relative horizontal clinical attachment level) | baseline to 9 months
change in probing depth | baseline to 9 months
change in site specific plaque index | baseline to 9 months
change in modified sulcus bleeding index | baseline to 9 months